CLINICAL TRIAL: NCT04790318
Title: Trans-incisional Quadratus Lumborum Block Versus Caudal Analgesia in Pediatric Open Renal Surgeries, a Randomized Clinical Trial.
Brief Title: Trans-incisional Quadratus Lumborum Block Versus Caudal Analgesia in Pediatric Open Renal Surgeries.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Amin Mohammed Alansary Amin Ahmed Helwa, Assistant professor, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: FMASU R 48/2020/2021
Record Dates: First submitted 2021-03-02; First posted 2021-03-10 (Actual); Last update posted 2022-12-21 (Actual); Status verified 2022-12

CONDITIONS: Anesthesia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- General Anesthesia +TiQLB (Active Comparator): patients will receive combined general anesthesia and quadratus lumborum block (trans-incisional) with 0.5 mL/kg of bupivacaine 0.2 %. with maximum volume limited to 20 ml
  Interventions: Procedure: Trans-incisional Quadratus lumborum block
- General Anesthesia+ Caudal block (Active Comparator): patients will receive combined general anesthesia and caudal analgesia (just after wound closure) with 1.25 mL/kg of bupivacaine 0.2 % (three parts 0.25 % bupivacaine to one part saline.
  Interventions: Procedure: Caudal block

INTERVENTIONS:
Procedure: Trans-incisional Quadratus lumborum block — patients will receive combined general anesthesia and quadratus lumborum block (trans-incisional) with 0.5 mL/kg of bupivacaine 0.2 %. with maximum volume was limited to 20 ml
  Arms: General Anesthesia +TiQLB
Procedure: Caudal block — patients will receive combined general anesthesia and caudal analgesia (just after wound closure) with 1.25 mL/kg of bupivacaine 0.2 % (three parts 0.25 % bupivacaine to one part saline.
  Arms: General Anesthesia+ Caudal block

SUMMARY:
There is scare literature about the usage of QLB in pediatric population, particularly the trans-incisional approach. Hence, the purpose of this study is to compare the postoperative analgesic efficacy of ultrasound-guided caudal epidural block versus ultrasound-guided QLB (trans-incisional) in combination with general anesthesia in pediatric patients undergoing elective open renal surgeries regarding pain scores, total analgesic consumption, and adverse effects.

ELIGIBILITY:
Inclusion Criteria:

1. patients who will be scheduled for indicated open pediatric renal surgery in the lateral decubitus position (nephrectomy, partial nephrectomy, pyeloplasty and nephrolithotomy for complex renal stones).
2. physical status American Society of Anesthesiologists (ASA) I or II.

Exclusion Criteria:

1. - patients whose guardians refuse to participate.
2. -ASA physical status >II. 3-patients who have contraindications to regional analgesic procedures. 4-patients who have major illnesses (e.g., cardiac, respiratory, renal, hepatic or neurological).

5-spine or chest wall deformity. 6-History of previous renal surgeries. 7-Coagulation abnormalities. 8-Infection at the injection site. 9-An allergy or contraindications to the drugs used in the study.

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2021-03-15 (Actual); Primary Completion 2022-09-15 (Actual); Study Completion 2022-10-20 (Actual)

PRIMARY OUTCOMES:
First time to analgesic requirement | 1st 24 hour
  Ketorolac is an IV NSAID that has been shown to have similar efficacy to morphine . Ketorolac will be dosed at 0.5 mg/kg every 6-8 hours for the 1st 24 h postoperatively as an analgesic after request.

SECONDARY OUTCOMES:
total analgesic consumption | 1st 24 hour
  Ketorolac will be dosed at 0.5 mg/kg every 6-8 hours for the 1st 24 h postoperatively as an analgesic after request.Total ketorolac consumption per 24 h will be calculated .
Face, leg, activity, cry, consolability scale (FLACC) | 1st 24 hours postoperatively
  Pain scores will be evaluated by a blinded observer anesthesiologist at the time of arrival in the PACU and 10, 20, and 30 min and 1, 2, 4, 6, 12, and 24 h thereafter using the face, leg, activity, cry, consolability scale (FLACC) (ranging from 0-10, where 0 = no pain, 10 = worst pain).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University hospitals, Cairo, Egypt